CLINICAL TRIAL: NCT05177159
Title: Postoperative Delirium and Its Biomarkers in Elderly Patients Undergoing Non-cardiac and Non-neurosurgery: a Prospective Cohort Study.
Brief Title: Postoperative Delirium and Its Biomarkers in Elderly Patients Undergoing Non-cardiac and Non-neurosurgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Other Study IDs: 2018-5-30
Record Dates: First submitted 2018-06-04; First posted 2022-01-04 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative delirium
  Interventions: Other: The regional cerebral oxygen saturation (rSO2); Other: The glial fibrillary acidic protein (GFAP); Other: The brain-derived-neurotrophic factor (BDNF)
- Non postoperative delirium
  Interventions: Other: The regional cerebral oxygen saturation (rSO2); Other: The glial fibrillary acidic protein (GFAP); Other: The brain-derived-neurotrophic factor (BDNF)

INTERVENTIONS:
Other: The regional cerebral oxygen saturation (rSO2) — Measurement of rSO2 with non-invasive near-infrared light spectrum monitor. The average, left and right frontal regions absolute rSO2 values will be collected every 30 seconds during the whole surgery until postoperative 2 hours, and the mean values will be calculated. Absolute rSO2 value and AUT (area under the threshold) send beneath the absolute threshold limits of 40%, 50% and 20%, 30% under the baseline. AUT will be calculated based on this formula: AUT (present)=AUT (past)+(rSO2 threshold-rSO2 value)×sample rate
Other: The glial fibrillary acidic protein (GFAP) — Venous blood sample will be collected and tested for plasma GFAP. The blood will be collected 10 minutes before anesthesia, 30 minutes after intubation, every hour during operation, 15 minutes after extubation, and at 10:00 AM in postoperative 1,3,5 days.
Other: The brain-derived-neurotrophic factor (BDNF) — Venous blood sample will be collected and tested for plasma BDNF. The blood will be collected 10 minutes before anesthesia, 30 minutes after intubation, every hour during operation, 15 minutes after extubation, and at 10:00 AM in postoperative 1,3,5 days.

SUMMARY:
Postoperative delirium (POD) is a common complication in elderly patients and is associated with negative clinical outcomes, such as prolonged hospitalizations, cognitive impairment, and higher mortality rate. While the pathophysiology of delirium remains unknown, the cerebral hypoperfusion and neuroinflammatory response are considered to play an important role in the process of POD. The aim of the study is to determine the association between POD and biomarkers in elderly patients undergoing noncardiac and non-neurological surgery.

ELIGIBILITY:
Inclusion Criteria:

* With American Society of Anesthesiologists (ASA) physical status Ⅱ-Ⅳ
* Undergo elective non-cardiac and non-neurological surgery receiving general anesthesia
* Operation time is expected to be longer than 2 hours

Exclusion Criteria:

* Clinical diagnosis of dementia
* Clinical diagnosis of cerebrovascular disorders
* Clinical diagnosis of heart failure
* Clinical diagnosis of liver failure
* Clinical diagnosis of renal failure
* Clinical diagnosis of traumatic brain injury
* Alcohol abuse
* Can not complete the cognitive assessments
* Refuse to sign informed consent

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients who schedule to receive elective non-cardiac and non-neurological surgery in Beijing Tiantan Hospital.
Sampling Method: Probability Sample
Enrollment: 417 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium within postoperative 5 days | the incidence of delirum within postoperative 5 days.
  The postoperative delirium will be diagnosed if patients have fluctuation in mental status and attention and either thinking or consciousness in the past 24 hours as evidenced by fluctuation on Confusion Assessment Method-Intensive Care Unit (CAM-ICU) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China